CLINICAL TRIAL: NCT05201248
Title: Phase 1b/2, Open-Label Trial to Evaluate Safety and Preliminary Efficacy of Epcoritamab As Monotherapy or Combined With Standard-of-Care Therapies in Chinese Subjects With B-Cell Non-Hodgkin Lymphoma
Brief Title: A Study to Evaluate Adverse Events and Change in Disease Activity of Subcutaneous (SC) Epcoritamab As Monotherapy or Combined With Standard of Care Therapies in Adult Participants in China With B-Cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M21-103
Record Dates: First submitted 2022-01-18; First posted 2022-01-21 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: B-Cell Non-Hodgkin Lymphoma
Keywords: B-Cell Non-Hodgkin Lymphoma; Epcoritamab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; R-CHOP; Rituximab; Lenalidomide; R2; ABBV-GMAB-3013; Cancer; EPCORE
MeSH Terms: conditions — Lymphoma, B-Cell; Neoplasms | interventions — Cyclophosphamide; Rituximab; Doxorubicin; Vincristine; Prednisone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 Part 1: Epcoritamab Monotherapy (Experimental): Participants will receive subcutaneous (SC) epcoritamab in 28 day cycles.
  Interventions: Drug: Epcoritamab
- Cohort 1 Part 2: Epcoritamab Expansion (Experimental): Participants will receive SC epcoritamab in 28 day cycles.
  Interventions: Drug: Epcoritamab
- Cohort 2: Epcoritamab + RCHOP (Experimental): Participants will receive SC epcoritamab in combination with [intravenously (IV) infused rituximab, IV injected cyclophosphamide, IV infused doxorubicin, IV infused vincristine, and oral prednisone (R-CHOP)] in 21 day cycles followed by 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- Cohort 3: Epcoritamab + R2 (Experimental): Participants will receive SC epcoritamab in combination with [intravenously (IV) infused rituximab, and oral lenalidomide (R2)] in 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Epcoritamab — Subcutaneous Injection (SC)
  Other Names: ABBV-GMAB-3013
Drug: Cyclophosphamide — IV Injection
  Arms: Cohort 2: Epcoritamab + RCHOP
Drug: Rituximab — Intravenous (IV) Infusion
  Arms: Cohort 2: Epcoritamab + RCHOP; Cohort 3: Epcoritamab + R2
Drug: Doxorubicin — IV Infusion
  Arms: Cohort 2: Epcoritamab + RCHOP
Drug: Vincristine — IV Infusion
  Arms: Cohort 2: Epcoritamab + RCHOP
Drug: Prednisone — Oral; Tablet
  Arms: Cohort 2: Epcoritamab + RCHOP
Drug: Lenalidomide — Oral; Capsule
  Arms: Cohort 3: Epcoritamab + R2

SUMMARY:
B-cell Lymphoma is an aggressive and rare cancer of a type of immune cells (a white blood cell responsible for fighting infections). The purpose of this study is to assess the safety and toxicity of epcoritamab as a monotherapy and when combined with standard of care therapy [Rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) or Rituximab and lenalidomide (R2)] in adult participants in China with B-Cell Non-Hodgkin Lymphoma. Adverse events and change in disease activity will be assessed.

Epcoritamab is an investigational drug being developed for the treatment of B-Cell Non-Hodgkin Lymphoma. Study doctors put the participants in groups called treatment arms. A monotherapy of epcoritamab and two different combination of epcoritamab with standard of care therapy (R-CHOP or R2) will be explored. Each treatment arm receives a different treatment combination depending on stage of the study and eligibility. Approximately 66 adult participants with B-Cell Non-Hodgkin Lymphoma will be enrolled in the study in approximately 21 sites in China.

In the monotherapy arm (Cohort 1), participants will receive subcutaneous epcoritamab in 28-day cycles. In the combination arms (Cohorts 2 and 3), participants in Cohort 2 will receive subcutaneous epcoritamab with standard of care therapy (R-CHOP) in 21-day cycles followed by 28-day cycles, participants in Cohort 3 will receive subcutaneous epcoritamab with standard of care therapy (R2) in 28-day cycles.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

All Cohorts:

* Life expectancy of >= 3 months on standard of care (SOC).
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status score 0 - 2.
* Has one or more measurable disease sites:

  * Fluorodeoxyglucose-positron emission tomography (FDGPET) scan demonstrating positive lesion compatible with computed tomography (CT) or magnetic resonance image (MRI)-defined anatomical tumor sites.
  * >= 1 measurable nodal lesion (long axis > 1.5 cm and short axis > 1.0 cm) or >= 1.0 measurable extra-nodal lesion (long axis >= 1 cm) on CT scan or MRI. Note: A previously irradiated lesion must have demonstrated progression or residual disease in the lesion after radiotherapy to be considered measurable.

Cohort 1 Part 1 (Monotherapy Safety Run-in) Specific Criteria:

* Must have histologically confirmed CD20+ Diffuse large B-cell lymphoma (DLBCL), or High-grade B-cell lymphoma (HGCBL) with MYC and BCL2 and/or BCL6 translocations and DLBCL feature, and follicular Lymphoma (FL) at most recent (previous or current) representative tumor biopsy based on the pathology report, according to the World Health Organization (WHO) 2016 (or later) classification.
* Must have at least one prior treatment with an anti-CD20 monoclonal antibody (e.g., rituximab) potentially in combination with chemotherapy and/or relapsed after autologous stem cell rescue.
* Must have relapsed or refractory disease. Note: Relapsed disease is defined as disease that has recurred >= 6 months after completion of therapy. Refractory disease is defined as disease that either progressed or failed to achieve an objective response during therapy or progressed within 6 months (<6 months) of completion of therapy.

Cohort 1 Part 2 (Monotherapy Expansion) Specific Criteria:

* Must have histologically confirmed CD20+ DLBCL at most recent (previous or current) representative tumor biopsy based on the pathology report, inclusive of the following according to the World Health Organization (WHO) 2016 (or later) classification.

  * DLBCL, not otherwise specified (NOS) including de novo or histologically transformed from an earlier diagnosis of indolent lymphoma such as FL and nodal marginal zone lymphoma with a subsequent development of DLBCL relapse or.
  * "Double-hit" or "triple-hit" with DLBCL morphology (technically classified in WHO 2016 as HGBCL, with MYC and BCL2 and/or BCL6 translocations). Note: Double- /triple-hit lymphomas without DLBCL morphology and those classified in WHO 2016 as HGBCL, NOS are not eligible.
  * FL Grade 3B.
* Following safety run-in and up to the 12th participant (including the number of safety run-in participants) in Cohort 1, participants must have received at least 1 prior line of systemic therapies which must include an anti-CD20 monoclonal antibody containing combination therapy (e.g., rituximab). After safety run-in confirms tolerability of the full dose A of epcoritamab, participants must have received at least 2 prior lines of systemic therapies.
* Must have either failed prior autologous HSCT, or be ineligible for autologous HSCT due to age, comorbidities, performance status, comorbidities, or insufficient response to prior treatment.
* Must have relapsed or refractory disease. Note: Relapsed disease is defined as disease that has recurred >= 6 months after completion of therapy. Refractory disease is defined as disease that either progressed or failed to achieve an objective response during therapy or progressed within 6 months (< 6 months) of completion of therapy.

Cohort 2 Specific Criteria:

* Must have newly diagnosed CD20+ DLBCL.
* Must have one of the following histologically confirmed CD20+ DLBCL (de novo or histologically transformed from FL at most recent (previous or current) representative tumor biopsy based on the pathology report including one of the following diagnoses according to the WHO 2016 (or later) classification:

  * DLBCL, not otherwise specified (NOS);
  * "Double-hit" or "triple-hit" with DLBCL morphology (technically classified in WHO 2016 as HGBCL, with MYC and BCL2 and/or BCL6 translocations) Note: Double-/triple-hit lymphomas without DLBCL morphology and those classified in WHO 2016 as HGBCL, NOS are not eligible or;
  * FL Grade 3B
* Eligible for standard R-CHOP for 6 cycles.

Cohort 3 Specific Criteria:

* Must have histologically confirmed CD20+ Grade 1 - 3a Follicular Lymphoma stage II, III, or IV with no evidence of histologic transformation to an aggressive lymphoma at most recent (previous or current) representative tumor biopsy and based on the pathology report, according to the WHO 2016 (or later) classification.
* Must have R/R disease to at least one prior systemic anti-lymphoma treatment which must include an anti CD20 monoclonal antibody (e.g., rituximab). Participant who received only prior anti-CD20 monoclonal antibody monotherapy is not eligible. Note: Relapsed disease is defined as disease that previously responded to therapy but progressed >= 6 months after completion of therapy. Refractory disease is defined as disease that either progressed during therapy, failed to achieve an objective response or progressed within 6 months (< 6 months) of completion of therapy.
* Must be eligible for R2 per investigator determination.
* Willing to take aspirin prophylaxis (participants with low or intermediate risk for thromboembolism) or prophylactic anticoagulant (if high risk for a thromboembolic event) (lenalidomide treated participants only).

Exclusion Criteria:

All Cohorts:

* History of primary mediastinal lymphoma.
* Autologous Stem Cell Transplantation within 100 days prior to enrollment.
* Have received prior allogeneic hematopoietic stem cell transplantation at any time.
* Have been treated with a bispecific antibody targeting CD3 and CD20.

Cohort 2 Specific Criteria:

- History of prior systemic anti-lymphoma therapy (including definitive radiotherapy) for Diffuse large B-cell lymphoma (DLBCL) other than corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 Part 2 [(3L+) R/R DLBCL]: Best Overall Response (BOR) | Up to Approximately 5 Years
  Best overall response (BOR) is defined as the percentage of participants in Cohort 1 Part 2 third line plus (3L) R/R DLBCL who achieved best overall response of complete response (CR) or partial response (PR) by Lugano 2014 criteria as assessed by independent review committee (IRC).
Cohort 1 Part 1, Cohort 2, and Cohort 3: Number of Incidence of Dose-Limiting Toxicities (DLT) | Up to Approximately 5 Years
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.

SECONDARY OUTCOMES:
Cohort 1 Part 2 [(3L+) R/R DLBCL]: Percentage of Participants with Complete Remission (CR) | Up to Approximately 5 Years
  CR is defined as the absence of lymphoma determined by Lugano 2014 criteria as assessed by IRC.
Cohort 1 Part 2 [(3L+) R/R DLBCL]: Number of Participants with Progression-free survival (PFS) | Up to Approximately 5 Years
  PFS is defined as the time in months from the first dose of study drug to the earliest occurrence of radiographic progression determined by Lugano 2014 criteria as assessed by IRC, or death from any cause.
Cohort 1 Part 2 [(3L+) R/R DLBCL]: Overall survival (OS) | Up to Approximately 5 Years
  OS is defined for Cohort 1 epcoritamab monotherapy participants, as the time in months from first dose of epcoritamab to death from any cause.
Cohort 1 Part 2 [(3L+) R/R DLBCL]: Duration of response (DOR) | Up to Approximately 5 Years
  DOR is defined for participants who achieved best overall response of CR or PR ('responders'), as the time in months from initial CR/PR to the earliest occurrence of radiographic progression determined by Lugano 2014 criteria as assessed by IRC, or death from any cause.
Cohort 1 Part 2 [(3L+) R/R DLBCL]: Time-to-response (TTR) | Up to Approximately 5 Years
  TTR is defined as the number of months from the date of first dose to the date of best overall response of CR or PR ('responders') determined by Lugano 2014 criteria as assessed by IRC.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (18):
- China (18):
  - The Fifth Medical Center of PLA General Hospital /ID# 230520, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 228138, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital /ID# 231890, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center /ID# 228033, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital /ID# 228028, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 227916, Guangzhou, Guangdong
  - Henan Cancer Hospital /ID# 228772, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Sc /ID# 231221, Wuhan, Hubei
  - Hunan Cancer Hospital /ID# 231859, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University /ID# 228024, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College /ID# 228774, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 228771, Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital /ID# 231944, Nanchang, Jiangxi
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 227724, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 231434, Chengdu, Sichuan
  - Tianjin Cancer Hospital /ID# 228135, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 228154, Hangzhou, Zhejiang
  - Zhejiang Cancer hospital /ID# 228776, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/